CLINICAL TRIAL: NCT05738733
Title: A Proof of Science, In-Use Tolerance, Safety, and Efficacy Clinical Study of MsChief Personal Lubricant in Healthy Female Subjects
Brief Title: A Clinical Efficacy Study of MsChief Personal Lubricant in Healthy Female Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: TTK Healthcare Ltd - Protective Devices Division (Unknown)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator - Medical Director, NovoBliss Research Pvt Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NB230002-TT
Record Dates: First submitted 2023-01-31; First posted 2023-02-22 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Healthy Females

STUDY DESIGN:
Intervention Model Description: A proof-of-science, open-label, single-centre, four-arm, In-Use tolerance, safety, efficacy clinical study
Masking Description: The study is open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MsChief Classic Natural Lubricant (Experimental): MsChief Classic natural lubricant contains aqua, propylene glycol, hydroxyethyl cellulose, ethyl menthane carboxamide and methyl diisopropyl propionamide, aloe barbadensis leaf juice, benzoic acid, hippophae Rhamnoides extract, tocophersolan, sodium hydroxide. MsChief Classic natural lubricant is a special moisturizer with aloe vera, vitamin E and sea buckthorn. It not only conditions but also moisturises the skin. This lubricant is water-based is free of sugar or saccharine. This product does not contain paraben or glycerine. This product has a unique formulation pH ideal for intimate area.
  Interventions: Device: MsChief Classic Natural Lubricant
- MsChief Ylang Ylang Natural Lubricant (Experimental): MsChief Ylang Ylang natural lubricant contains aqua, propylene glycol, flavour, hydroxyethyl cellulose, ethyl menthane carboxamide and methyl diisopropyl propionamide, aloe barbadensis leaf juice, benzoic acid, hippophae Rhamnoides extract, tocophersolan, sodium hydroxide. MsChief Ylang Ylang natural lubricant is a special moisturizer with aloe vera, vitamin E and sea buckthorn It not only conditions but also moisturise the skin. This lubricant is water-based contain natural flavour and free of sugar or saccharine. This product does not contain paraben or glycerine. This product has a unique formulation pH ideal for intimate area.
  Interventions: Device: MsChief Ylang Ylang Natural Lubricant
- MsChief Vanilla & Citrus Natural Lubricant (Experimental): MsChief vanilla and citrus natural lubricant contain aqua, propylene glycol, flavour, hydroxyethyl cellulose, ethyl menthane carboxamide and methyl diisopropyl propionamide, aloe barbadensis leaf juice, benzoic acid, hippophae Rhamnoides extract, tocophersolan, sodium hydroxide. MsChief vanilla and citrus natural lubricant is a special moisturizer with Aloe vera, vitamin E and sea buckthorn. It not only conditions but also moisturise the skin. This lubricant is water based contain natural flavour and free of sugar or saccharine. This product does not contain paraben or glycerine. This product has a unique formulation pH ideal for intimate area.
  Interventions: Device: MsChief Vanilla & Citrus Natural Lubricant
- MsChief Tea & Peach Natural Lubricant (Experimental): MsChief tea & peach natural lubricant contains aqua, propylene glycol, flavour, hydroxyethyl cellulose, ethyl menthane carboxamide and methyl diisopropyl propionamide, aloe barbadensis leaf juice, benzoic acid, hippophae Rhamnoides extract, tocophersolan, sodium hydroxide. MsChief tea & peach natural lubricant is a special moisturizer with Aloe vera, vitamin E and sea buckthorn. It not only conditions but also moisturises the skin. This lubricant is water-based contains natural flavour and is free of sugar or saccharine. This product does not contain paraben or glycerine. This product has a unique formulation pH ideal for intimate area.
  Interventions: Device: MsChief Tea & Peach Natural Lubricant

INTERVENTIONS:
Device: MsChief Classic Natural Lubricant — Apply the desire amount of lubricant on the body to make it more sensitive.
  Arms: MsChief Classic Natural Lubricant
Device: MsChief Ylang Ylang Natural Lubricant — Apply the desire amount of lubricant on the body to make it more sensitive.
  Arms: MsChief Ylang Ylang Natural Lubricant
Device: MsChief Vanilla & Citrus Natural Lubricant — Apply the desire amount of lubricant on the body to make it more sensitive.
  Arms: MsChief Vanilla & Citrus Natural Lubricant
Device: MsChief Tea & Peach Natural Lubricant — Apply the desire amount of lubricant on the body to make it more sensitive.
  Arms: MsChief Tea & Peach Natural Lubricant

SUMMARY:
A Proof of Science, Open-Label, Single Centre, Four-Arm, In-Use Tolerance, Safety, and Efficacy Clinical Study of MsChief Personal Lubricant in Healthy Female Subjects.

30 subjects/product (33 subjects' enrolment/treatment) healthy non-pregnant/non-lactating females with an age of 18 - 65 years old.

A total of up to 132 subjects (33 subjects/product) will be enrolled to get 120 completed subjects (30 subjects/product) in the study.

DETAILED DESCRIPTION:
A sufficient number of healthy female subjects with an age group of 18 - 65 years old with a Nugent score ≤3 will be recruited/enrolled.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. The subjects will be instructed to visit the facility as per the below visits

* Visit 01 (Within 07 Days): Screening, Baseline evaluations
* Visit 02 (Day 01): Enrolment & Test Products usage phase start
* Visit 03 (Day 16): Test Products usage ends, End of the study Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be telephonically contacted by recruiting department prior to the enrolment visit. Subjects will be instructed during screening (prior to enrolment) not to use any other product for intimate washes, lubricant, or any other product during the study.

Assessment of efficacy parameters will be done before test products usage on Day 1 and will be compared with after test products usage during Day 16 as listed below.

1. Gynaecological Assessments

   * Local irritation, pruritus, erythema, edema
   * Moisturizing effect - moisture, dryness, flaking, epithelial mucosa
   * Quality and odour of vaginal discharge
   * Vaginal pH measure using pH paper
   * Clinical symptoms associated with infections
   * Verbal rating scale (0-4 score)- Vaginal itching
2. Subjective Self-assessments

   * Perceived irritations - Burning, Itching, Stinging, Discomfort
   * Sexual activity (where appropriate)
   * VAS Scoring for Vaginal itchiness
   * Quality of life assessment
3. Microbiological Assessments • Nugents scoring

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years (both inclusive) at the time of consent.
2. Sex: Healthy non-pregnant/non-lactating females

   * Females of fertile reproductive age with a propensity to vulvo-vaginal infection (18 years to 40 years)
   * Females in the pre-menopausal age group (41 years to 48 years)
   * Females in the post-menopausal age group (49 years to 65 years)
3. The subject is with Nugent score ≤3.
4. The subject with an active sex life of at least 01 sexual intercourse in a week
5. The subject of childbearing potential must have a reported negative pregnancy during screening and the end of the study.
6. The subject without a history of sensitivity to similar products/formulations
7. The subject is willing to give written informed consent and is willing to follow the study procedures.
8. The subject is willing to abide by the study protocol and study restrictions including abstinence from the use of any other product besides the test product for intimate wash, lubricant or any other products during the study.
9. The subject is a personal lubricant user and agrees to replace her usual personal lubricant with the test product.
10. The subject of childbearing potential who is willing to use a highly effective method of contraception throughout the clinical investigation.
11. The subject is of childbearing potential, is practising and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
12. If currently using hormonal contraception, has been using this form of contraception for at least 6 months and agrees to continue using the same contraception for the duration of the study.
13. The subject who agrees to have a gynaecological pelvic examination to ensure no significant disease findings and have intact skin and mucous in the test region assessed by the gynaecologist at all the relevant time points

Exclusion Criteria:

1. The subject used other intra-vaginal gel moisturizers during the study.
2. The subject with Nugent score >3.
3. The subject who is diagnosed with cancer
4. The subject using hormone replacement therapy for the last 3 months
5. The subject has a history or visible evidence of chronic skin disease or regional infections, genital herpes, vaginal infections or urinary tract infections.
6. Pregnant or lactating, women who are likely to become pregnant.
7. The subject exhibits or reports gynecologic abnormalities or has had vaginitis within 60 days prior to study initiation.
8. Personal history of allergy and hypersensitivity to any product of feminine hygiene, severe systemic complications of viral infections, severe systemic illness like cardiovascular disorders, neurological disorders, renal disorders, and autoimmune disorders.
9. The subject with any form of chronic infection/ allergy/ disease which may influence the study result
10. The subject with bacterial vaginosis/candidiasis/mycotic infections
11. The subject participated in clinical studies or had received any investigational agent in the previous 30 days.
12. The subject is not willing to sign an informed consent form.
13. The subject is an employee at the site or a partner or first-degree relative of the Investigator.
14. The subject fails to satisfy the Investigator of fitness to participate for any other reason.
15. The subject has had previous episodes of vaginal bleeding of unknown origin within the last 6 months of the screening visit.
16. The subject showed vaginal prolapse and/or other medical conditions that could interfere with the study's conduct and participation.
17. The subject who has used any kind of systemic and/or local hormonal products for vaginal dryness or any other vaginal condition in the 3 months prior to screening

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change in vaginal local irritation | From baseline i.e. Day 01 (before application) to Day 16 post usage
  To assess the test product(s) effectiveness in terms of change in vaginal local irritation by the Gynecologist using 4-point scale[0=absent, 1=mild, 2=moderate, 3=severe]..
Change in vaginal moisturizing effects | From baseline i.e. Day 01 (before application) to Day 16 post usage
  To assess the test product(s) effectiveness in terms of change in vaginal moisturizing effects as evaluated by the Gynecologist using Modified Schemer Test
Change in sexual intimacy | From baseline i.e. Day 01 (before application) to Day 16 post usage
  To assess the test product(s) effectiveness in terms of change in sexual intimacy using female sexual function index self-reported scale score [score of zero indicates that the subject reported having no sexual activity during the past 15 days].
Change in VAS score for vaginal itching | From baseline i.e. Day 01 (before application) to Day 16 post usage
  To assess the test product(s) effectiveness in terms of change in Visual Analog Score score for vaginal itching as evaluated by the Gynecologist [ 0 points - No itchiness, greater than or equal to 9 points: Very severe Itchiness

SECONDARY OUTCOMES:
Change in quality and odor of vaginal discharge | From baseline i.e. Day 01 (before application) to Day 16 post usage
  To assess the test product(s) effectiveness in terms of change in quality and odor of vaginal discharge as evaluated by the Gynecologist using vaginal odour score [0=absent, 1=mild, 2=moderate, 3=intense, 4=very intense].
Change in vaginal pH | From baseline i.e. Day 01 (before application) to Day 16 post usage
  To assess the test product(s) effectiveness in terms of change in vaginal pH as evaluated by the Gynecologist using pH paper
Change in clinical symptoms associated with infection | From baseline i.e. Day 01 (before application) to Day 16 post usage
  To assess the test product(s) effectiveness in terms of change in clinical symptoms associated with infection i.e. redness, itching, burning sensation, swelling of vaginal vulva, vaginal rash as evaluated by the Gynecologist using 4-point scale [0=absent, 1=mild, 2=moderate, 3=severe].
Change in Nugents score | From baseline i.e. Day 01 (before application) to Day 16 post usage
  To assess the test product(s) effectiveness for change in Nugents score for microbial assessment [0-3: Normal, 4-6: Intermediate bacterial count, 7-10: Bacterial vaginosis].
Product perception and consumer feedback | From baseline i.e. Day 01 (before application) to Day 16 post usage
  To assess the effect of the test product(s) assessed in terms of product perception and consumer feedback using 9 point hedonic scoring scale

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nayan K Patel, MBBS, Principal Investigator — Medical Director
Locations (1):
- Krisha Hospital, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No